CLINICAL TRIAL: NCT00998140
Title: Optimizing Resuscitation After Cardiac Arrest in the Community: Increasing the Probability of Survival While Reducing Costs
Brief Title: Optimizing Resuscitation After Cardiac Arrest in the Community
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr Sharon Einav, Dr., Shaare Zedek Medical Center
Other Study IDs: NIHPR 08/90/a
Record Dates: First submitted 2009-10-18; First posted 2009-10-20 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Cardiopulmonary Arrest Outcome
Keywords: resuscitation; sudden death; cardiopulmonary resuscitation; emergency medical services; termination of resuscitation; ventricular fibrillation; out-of-hospital cardiac arrest; asystole; medical futility; withdrawing treatment; transportation of patients; health expenditures; healthcare costs
MeSH Terms: conditions — Death, Sudden; Ventricular Fibrillation; Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Resuscitative efforts have been shown to be unsuccessful in most cases of out-of-hospital cardiac arrest (OHCA), and survivors who do recover cardiac function often sustain severe hypoxic brain damage. Time to efficacious care is a primary determinant of disability-free survival. In the Jerusalem district, only 9% of OHCA patients present with ventricular tachycardia/ventricular fibrillation (VT/VF) as the primary rhythm, whereas 77% present with asystole; this seems primarily to be the result of long collapse-to-arrival times. Nevertheless, overly zealous resuscitation is undertaken in a high proportion of arrests with a futile prognosis, leading to excessive costs.

Study hypotheses:

1. Subpopulations for whom intervention is futile/counter-productive are identifiable
2. Substantial waste of resources can be avoided
3. Optimization of emergency medical services (EMS) reorganization without adding resources is an achievable goal

ELIGIBILITY:
Inclusion Criteria:

* All victims of non-traumatic out-of hospital cardiopulmonary arrest (defined as the absence of either spontaneous respiration or palpable pulse or both) within the Jerusalem district.

Exclusion Criteria:

* Patients with do-not-resuscitate orders or an advance directive to that effect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All victims of non-traumatic out-of hospital cardiopulmonary arrest (defined as the absence of either spontaneous respiration or palpable pulse or both) within the Jerusalem district.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2009-03; Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Einav, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Pachys G, Kaufman N, Bdolah-Abram T, Kark JD, Einav S. Predictors of long-term survival after out-of-hospital cardiac arrest: the impact of Activities of Daily Living and Cerebral Performance Category scores. Resuscitation. 2014 Aug;85(8):1052-8. doi: 10.1016/j.resuscitation.2014.03.312. Epub 2014 Apr 12. PMID 24727137